CLINICAL TRIAL: NCT05418855
Title: Clinical Characteristics and Outcomes of SLE Patients Admitted to Assiut University Hospital Critical Care Unit
Brief Title: Clinical Characteristics and Outcomes of SLE Patients Admitted to Critical Care Unit
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, MOHussein, Resident doctor at critical care unit of internal medicine department at Assiut University Hospitals, Assiut University
Other Study IDs: SLE Patients in CCU.
Record Dates: First submitted 2022-02-04; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present work is to determine the frequency of critical complications of SLE patients admitted to the intensive care unit,study the risk factors and out comes.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a systemic heterogeneous autoimmune disease with a highly variable course and prognosis that many different organs may be affected . It has wide spectrum of clinical presentation that affects all ages and ethnicities . Child-bearing women most often afflicted by this diseases, but with different disease manifestations and with variable severity .

The pathogenesis of SLE is complex and still largely unknown. Genetic, environmental, and hormonal factors contribute to disease susceptibility . The diagnosis of SLE is based on characteristic clinical findings of the skin, joints, kidneys, and the central nervous system, as well as on serological parameters such as antinuclear antibodies (ANA) . SLE mainly causes damage to the kidney, heart, joints, blood vessels, liver, lungs and the nervous system . Since SLE is a heterogeneous disease, its complications may vary and the severity or intensity depends on the area affected. Pulmonary hypertension, alveolar haemorrhage, thrombocytopenia, catastrophic antiphospholipid syndrome (APS), haemolytic anemia, neutropenia, blood cancer and thrombotic thrombocytopenic purpura, atherosclerosis, pericardial tamponade myocarditis, heart failure, arthritis, vasculitis, adrenal insufficiency, lupus nephritis (LN), neuropsychiatric disorders, pancreatitis, and myelitis are some of the major complications of SLE . In a previous study on Egyptian SLE patients, pleuro-pulmonary system was found to be one of the most commonly affected systems; pleurisy being the most frequent clinical finding followed by pulmonary infection and disease activity was an important predictor for infection .

Lupus flares and infections are the most common causes of admission to the ICU in patients with SLE. Pertaining to complications from infections, lower pulmonary tract infections are typically more severe and frequent.

A number of studies have addressed the characteristics and outcomes of critically ill SLE patients. In a cohort of 2870 SLE patients retrieved from a national database, the leading causes of ICU admission were found to be infections and organ dysfunction (neurological, cardiovascular, and respiratory systems).

Ethnic differences, availability of therapy, and health-care referral systems may impact SLE manifestation and prognosis. Few studies have provided a clinical characterization of SLE patients admitted to the ICU, and data on predictors of patient outcomes are discordant.

ELIGIBILITY:
Inclusion Criteria:

* SLE Patients Admitted to ICU.

Exclusion Criteria:

* Patients who stayed <48 h in ICU.
* Patients with major chronic organ disease not related to SLE or terminal cancer.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients fulfill the Systemic lupus international Collaborating Clinics (SLICC) Criteria for classification of SLE .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
complications of SLE patients admitted to the intensive care unit. | Baseline
  Number of incidence of complications depending on these measures will be reported Liver bilrubin alb Urea creatinine GFR CBC Ecg X Ray chest cardiomegaly effusion pulmonary edema Ct brain hge infarction Blood gases Clinical data Fever Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Bahy Ahmed, lecturer, Principal Investigator — Assiut University